CLINICAL TRIAL: NCT02590809
Title: Hypertrophic Cardiomyopathy Symptom Release by BX1514M
Acronym: Light-CARMIDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHUBX 2015/14
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2017-02

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Left ventricular obstruction
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): 20 patients
  Interventions: Drug: Treatment BX1514M; Other: Walk distance test; Other: Exercise echocardiography
- Placebo group (Placebo Comparator): 20 patients
  Interventions: Drug: Placebo; Other: Walk distance test; Other: Exercise echocardiography

INTERVENTIONS:
Drug: Treatment BX1514M — X mg x 3 /day of BX1514M for 15 days. Dosage will be then adapted, depending on symptoms release and walk distance test results for another 15 days period.
  Arms: Treatment group
Drug: Placebo — Placebo will be given for 30 days
  Arms: Placebo group
Other: Walk distance test — Walk distance test during 6 minutes
Other: Exercise echocardiography

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is the most frequent genetic cardiac disease characterized by an asymmetric hypertrophic. In two third of patients, an obstruction to blood ejection is observed within the left ventricle which is named left ventricular outflow tract obstruction (LVOTO). This phenomenon can occur at rest or during exercise and is associated with symptoms such as dyspnea, dizziness or chest pain that can significantly limit day life adaptation. To now, medical or interventional treatments such as betablocacker, calcium blockers or septal alcoholisation or surgery present with a limited efficiency. Recent studies from investigators group revealed new concepts about the role of venous return to the LVOTO. Therefore the investigators hypothesis that BX1514M generating a venous vascular constriction, could improve symptoms of HCM patients by reducing LVOTO.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a typical or atypical hypertrophic cardiomyopathy (HCM) confirmed by imaging modalities (echo and MRI) and/or genetic tests or a relative history of HCM
* Left ventricular obstruction during exercise on treadmill (above 50 mmHg)
* Positive response to leg lifting test (obstruction reduction above 20 mmHg) at rest or in early recovery phase
* Daily symptoms as shortness of breath during exercise (NYHA2-3), non coronary chest pain, dizziness
* Correct ultrasound windows quality
* Sinus rhythm
* Optimal medical treatment
* For women, pregnancy test or contraception
* Written consent form obtained

Exclusion Criteria:

* Previous treatment by BX1514M
* Extra-cardiac pathology with life expectancy below than 1 year
* No capability of consent form written
* Pregnancy women
* Secondary hypertension hypertrophy, secondary valvular disease hypertrophy
* Permanent atrial fibrillation
* Severe ventricular arrhythmia without Implantable Cardioverter Defibrillator (ICD)
* Severe coronary disease
* Severe non stabilized hypertension
* Severe cardiopathy (ejection fraction below 40% or demonstrated elevated end diastolic pressure or pulmonary pressure above 60 mmHg)
* Bradycardia
* Narrow angle glaucoma
* Vascular prethrombotic diseases
* Vascular spams
* Thyrotoxicosis
* Pheochromocytoma
* Severe renal failure (<30ml/mn)
* Patients at risk of urinary retention secondary to prostatic severe disease
* Raynaud's disease
* Non selective Monoamine Oxidase Inhibitors (MAOIs), iproniazid, nialamide or ephedrine, methylphenidate, phenylephrine, pseudoephedrine or digitalic
* Procedures modifying the peripheral venous return
* Participation to other research protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2016-07-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline at day 15 of covered distance during the 6 minutes walk distance test (6MWT) | Day 15
  In meters

SECONDARY OUTCOMES:
Covered distance during the 6 minutes walk distance test (6MWT) | Day 30
  In meters
Exercise echocardiography with measures of blood pressures in the rest and in the effort | Day 1, day 15, day 30

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane LAFITTE, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France